CLINICAL TRIAL: NCT03701321
Title: Phase 1/2 Study of Daratumumab, Bortezomib, Dexamethasone With or Without Venetoclax in Relapsed/Refractory Multiple Myeloma With Assessment for t(11;14) Status
Brief Title: Daratumumab, Bortezomib, and Dexamethasone With or Without Venetoclax in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02131; NCI-2018-02131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAA172 (Other: ECOG-ACRIN Cancer Research Group); U10CA180820 (NIH)
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; venetoclax

STUDY DESIGN:
Intervention Model Description: 3 arms in phase I, 2 arms in phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I (DVd, venetoclax) (Experimental): Patients receive daratumumab IV on days 1, 8, and 15 of cycles 1-3 and on day 1 of subsequent cycles, bortezomib SC on days 1, 8, and 15 of cycles 1-8, dexamethasone PO on days 1, 8, and 15 of cycles 1-8, and venetoclax PO QD on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Daratumumab; Drug: Dexamethasone; Drug: Venetoclax
- Phase II Arm D (DVd, venetoclax) (Experimental): Patients receive venetoclax PO QD on days 1-21, daratumumab IV on days 1, 8, and 15 of cycles 1-3 and on day 1 of subsequent cycles, bortezomib SC on days 1, 8, and 15 of cycles 1-8, and dexamethasone PO on days 1, 8, and 15 of cycles 1-8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Daratumumab; Drug: Dexamethasone; Drug: Venetoclax
- Phase II Arm E (DVd) (Active Comparator): Patients receive daratumumab IV on days 1, 8, and 15 of cycles 1-3 and on day 1 of subsequent cycles, bortezomib SC on days 1, 8, and 15 of cycles 1-8, and dexamethasone PO on days 1, 8, and 15 of cycles 1-8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
  Arms: Phase I (DVd, venetoclax); Phase II Arm D (DVd, venetoclax)

SUMMARY:
This phase I/II trial studies the side effects and best dose of venetoclax when given together with daratumumab, bortezomib, and dexamethasone, and how well they work in treating patients with multiple myeloma that has come back (relapsed) or does not respond to treatment (refractory). Drugs used in chemotherapy, such as venetoclax and dexamethasone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as daratumumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving venetoclax with daratumumab, bortezomib, and dexamethasone may work better in treating patients with relapsed or refractory multiple myeloma compared to standard of care treatment, including chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicities and the recommended phase II dose of venetoclax in combination with daratumumab, bortezomib, and dexamethasone for patients with relapsed/refractory multiple myeloma. (Phase I) II. To evaluate the safety of venetoclax (VEN) in combination with bortezomib and dexamethasone (DVd). (Phase I) III. To compare efficacy of DVd-VEN versus DVd as measured by minimal residual disease negative rate after 8 cycles of therapy. (Phase II) IV. To inform the role of t(11;14) as a biomarker in a subsequent evaluation of the regimen. (Phase II)

SECONDARY OBJECTIVES:

I. To compare rates of very good partial response between arms. II. To assess improvement in progression-free and overall survival with the addition of VEN.

III. To evaluate the safety of VEN in combination with DVd and compare overall toxicity rates between arms.

IV. To assess association of cycle 8 minimal residual disease (MRD) status with overall and progression-free survival.

V. To estimate the impact of t(11;14) status on very good partial response, overall and progression-free survival.

EXPLORATORY OBJECTIVES:

I. To measure treatment exposure and adherence. II. To estimate time to progression with the addition of VEN. III. To measure MRD levels longitudinally and assess the kinetics of relapse. IV. To assess association of MRD status after 8 cycles with survival outcomes. V. To evaluate agreement and discordance between methods determining disease-free status.

OUTLINE: This is a phase I, dose-escalation study of venetoclax followed by a phase II study.

PHASE I:

Patients receive daratumumab intravenously (IV) on days 1, 8, and 15 of cycles 1-3 and on day 1 of subsequent cycles, bortezomib subcutaneously (SC) on days 1, 8, and 15 of cycles 1-8, dexamethasone orally (PO) on days 1, 8, and 15 of cycles 1-8, and venetoclax PO once daily (QD) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM D: Patients receive venetoclax PO QD on days 1-21, daratumumab IV on days 1, 8, and 15 of cycles 1-3 and on day 1 of subsequent cycles, bortezomib SC on days 1, 8, and 15 of cycles 1-8, and dexamethasone PO on days 1, 8, and 15 of cycles 1-8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM E: Patients receive daratumumab IV on days 1, 8, and 15 of cycles 1-3 and on day 1 of subsequent cycles, bortezomib SC on days 1, 8, and 15 of cycles 1-8, and dexamethasone PO on days 1, 8, and 15 of cycles 1-8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I (ARMS A, B, C) - STEP 1: Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* PHASE I (ARMS A, B, C) - STEP 1: Patients must have been diagnosed with symptomatic relapsed/refractory multiple myeloma.

  * NOTE: Relapsed/refractory myeloma is defined as a disease which becomes non-responsive or progressive on therapy or within 60 days of the last treatment in patients who had achieved a minimal response (MR) or better on prior therapy.
* PHASE I (ARMS A, B, C) - STEP 1: t(11;14) status must be determined.
* PHASE I (ARMS A, B, C) - STEP 1: Patients must not have bortezomib refractory disease. Prior lenalidomide refractory patients are allowed.
* PHASE I (ARMS A, B, C) - STEP 1: Patients must have been treated with 1 or more lines of therapy. 1 prior line of systemic therapy is defined as 1 or more planned cycles of single agent or combination therapy, as well as a planned series of treatment regimens administered in a sequential manner (e.g. lenalidomide, bortezomib and dexamethasone induction therapy for 4 cycles followed by autologous stem cell transplantation and then lenalidomide maintenance therapy would be considered 1 line of prior therapy). Auto stem cell transplant is allowed provided the patient is 100 days out from stem cell infusion. Patients must not have had prior venetoclax. Allogeneic stem cell transplantation (SCT) patients are excluded.
* PHASE I (ARMS A, B, C) - STEP 1: Patients must have measurable disease as defined by having one or more of the following, obtained within 14 days prior to randomization:

  * >= 0.5 g/dL monoclonal protein (M-protein) on serum protein electrophoresis.
  * >= 200 mg/24 hrs of monoclonal protein (M-protein) on a 24 hour urine protein electrophoresis.
  * Involved free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio (< 0.26 or > 1.65).
* PHASE I (ARMS A, B, C) - STEP 1: Serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), and serum free light chain (FLC) assay are required to be performed within 14 days prior to randomization.

  * NOTE: UPEP (on a 24 hour collection) is required, no substitute method is acceptable. Urine must be followed monthly if the baseline urine M-spike is >= 200 mg/24 hr and urine in addition to serum must be followed in order to confirm a very good partial response (VGPR) or higher response.
  * NOTE: The serum free light chain test is required to be done if the patient does not have measurable disease in the serum or urine. Measurable disease in the serum is defined as having a serum M-spike >= 0.5 g/dL. Measurable disease in the urine is defined as having a urine M-spike >= 200 mg/24 hr.
* PHASE I (ARMS A, B, C) - STEP 1: Platelet count >= 100,000 cells/mm^3 (within 14 days prior to randomization).
* PHASE I (ARMS A, B, C) - STEP 1: Absolute neutrophil count >= 1000 cells/mm^3 (within 14 days prior to randomization).
* PHASE I (ARMS A, B, C) - STEP 1: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x the upper limit of normal (within 14 days prior to randomization).
* PHASE I (ARMS A, B, C) - STEP 1: Total bilirubin =< 1.5 x the upper limit of normal (within 14 days prior to randomization).
* PHASE I (ARMS A, B, C) - STEP 1: Calculated creatinine clearance >= 30 mL/min (within 14 days prior to randomization).
* PHASE I (ARMS A, B, C) - STEP 1: Hemoglobin >= 8.0 g/dL (within 14 days prior to randomization).
* PHASE I (ARMS A, B, C) - STEP 1: Women must not be pregnant or breast-feeding due to risk of fetal harm by the chemotherapeutic agents prescribed in this protocol. All females of childbearing potential must have a blood test or urine study within 7 days prior to registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* PHASE I (ARMS A, B, C) - STEP 1: Women of childbearing potential and sexually active males must use an accepted and highly effective method(s) of contraception or abstain from sexual intercourse for the duration of their participation in the study and for 3 months after the last dose of daratumumab or 30 days after the last dose of venetoclax, whichever is longer. Male patients must also agree not to donate sperm for the duration of their participation in the study for 3 months after the last dose of daratumumab or 30 days after the last dose of venetoclax whichever is longer.
* PHASE I (ARMS A, B, C) - STEP 1: Patients must not have > grade 2 neuropathy and/or a syndrome characterized by polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin change (POEMS).
* PHASE I (ARMS A, B, C) - STEP 1: Patients must not have New York Heart Association (NYHA) class III or IV heart failure or myocardial infarction within 6 months prior to registration.
* PHASE I (ARMS A, B, C) - STEP 1: Patients must avoid concomitant use of venetoclax with moderate or strong CYP3A inhibitors, strong or moderate CYP3A inducers, P-glycoprotein (P-gp) inhibitors, or narrow therapeutic index P-gp substrates.
* PHASE I (ARMS A, B, C) - STEP 1: Patients must not be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Patients with resolved infection (i.e., patients who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HepB) deoxyribonucleic acid (DNA) levels. Those who are PCR positive are not eligible. Patients with serologic findings suggestive of HepB vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HepB vaccination, do not need to be tested for HepB DNA by PCR. Patients with HepB core antibody (cAb) positive but HepB sAg negative, as well as HepB PCR negative, are eligible but will need to be monitored throughout the study.
* PHASE I (ARMS A, B, C) - STEP 1: Patients must not be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
* PHASE II (ARMS D, E) - STEP 1: ECOG performance status of 0-2.
* PHASE II (ARMS D, E) - STEP 1: Patients must have been diagnosed with symptomatic relapsed/refractory multiple myeloma.

  * NOTE: Relapsed/refractory myeloma is defined as a disease which becomes non-responsive or progressive on therapy or within 60 days of the last treatment in patients who had achieved a minimal response (MR) or better on prior therapy.
* PHASE II (ARMS D, E) - STEP 1: t(11;14) status must be determined.
* PHASE II (ARMS D, E) - STEP 1: Patients must not have bortezomib refractory disease. Prior lenalidomide refractory patients are allowed.
* PHASE II (ARMS D, E) - STEP 1: Patients must have been treated with 1 or more lines of therapy. 1 prior line of systemic therapy is defined as 1 or more planned cycles of single agent or combination therapy, as well as a planned series of treatment regimens administered in a sequential manner (e.g. lenalidomide, bortezomib and dexamethasone induction therapy for 4 cycles followed by autologous stem cell transplantation and then lenalidomide maintenance therapy would be considered 1 line of prior therapy). Auto stem cell transplant is allowed provided the patient is 100 days out from stem cell infusion. Patients must not have had prior venetoclax. Allogeneic SCT patients are excluded.
* PHASE II (ARMS D, E) - STEP 1: Patients must have measurable disease as defined by having one or more of the following, obtained within 14 days prior to randomization:

  * >= 0.5 g/dL monoclonal protein (M-protein) on serum protein electrophoresis.
  * >= 200 mg/24 hours (hrs) of monoclonal protein (M-protein) on a 24 hour urine protein electrophoresis.
  * Involved free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio (< 0.26 or > 1.65).
* PHASE II (ARMS D, E) - STEP 1: SPEP, UPEP, and serum FLC assay are required to be performed within 14 days prior to randomization.

  * NOTE: UPEP (on a 24 hour collection) is required, no substitute method is acceptable. Urine must be followed monthly if the baseline urine M-spike is >= 200 mg/24 hr. Please note that if both serum and urine m-components are present, both must be followed in order to evaluate response.
  * NOTE: The serum free light chain test is required to be done if the patient does not have measurable disease in the serum or urine. Measurable disease in the serum is defined as having a serum M-spike >= 0.5 g/dL. Measurable disease in the urine is defined as having a urine M-spike >= 200 mg/24 hr.
* PHASE II (ARMS D, E) - STEP 1: Platelet count >= 100,000 cells/mm^3 (within 14 days prior to randomization).
* PHASE II (ARMS D, E) - STEP 1: Absolute neutrophil count >= 1000 cells/mm^3 (within 14 days prior to randomization).
* PHASE II (ARMS D, E) - STEP 1: AST and ALT =< 2.5 x the upper limit of normal (within 14 days prior to randomization).
* PHASE II (ARMS D, E) - STEP 1: Total bilirubin =< 1.5 x the upper limit of normal (within 14 days prior to randomization).
* PHASE II (ARMS D, E) - STEP 1: Calculated creatinine clearance >= 30 mL/min (within 14 days prior to randomization).
* PHASE II (ARMS D, E) - STEP 1: Hemoglobin >= 8.0 g/dL (within 14 days prior to randomization).
* PHASE II (ARMS D, E) - STEP 1: Women must not be pregnant or breast-feeding due to risk of fetal harm by the chemotherapeutic agents prescribed in this protocol. All females of childbearing potential must have a blood test or urine study within 7 days prior to registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* PHASE II (ARMS D, E) - STEP 1: Women of childbearing potential and sexually active males must use an accepted and highly effective method(s) of contraception or abstain from sexual intercourse for the duration of their participation in the study and for 3 months after the last dose of daratumumab or 30 days after the last dose of venetoclax, whichever is longer. Male patients must also agree not to donate sperm for the duration of their participation in the study for 3 months after the last dose of daratumumab or 30 days after the last dose of venetoclax, whichever is longer.
* PHASE II (ARMS D, E) - STEP 1: Patients must not have > grade 2 neuropathy and/or POEMS.
* PHASE II (ARMS D, E) - STEP 1: Patients must not have NYHA Class III or IV heart failure or myocardial infarction within 6 months prior to registration.
* PHASE II (ARMS D, E) - STEP 1: Patients must avoid concomitant use of venetoclax with moderate or strong CYP3A inhibitors, strong or moderate CYP3A inducers, P-gp inhibitors, or narrow therapeutic index P-gp substrates.
* PHASE II (ARMS D, E) - STEP 1: Patients must not be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Patients with resolved infection (i.e., patients who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HepB) DNA levels. Those who are PCR positive are not eligible. Patients with serologic findings suggestive of HepB vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HepB vaccination, do not need to be tested for HepB DNA by PCR. Patients with HepB cAb positive but HepB sAg negative, as well as HepB PCR negative, are eligible but will need to be monitored throughout the study.
* PHASE II (ARMS D, E) - STEP 1: Patients must not be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy). However, patients who test negative for HepC by PCR may participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-25 (Estimated); Primary Completion 2020-05-28 (Estimated); Study Completion 2020-05-28 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of venetoclax in combination with daratumumab, bortezomib and dexamethasone (Phase I) | Up to 35 days
  Highest dose at which fewer than one-third of patients experience a dose-limiting toxicity.
Minimal residual disease (MRD) negative status (Phase II) | After cycle 8
  Per revised International Myeloma Working Group (IMWG) response criteria for next-generation sequencing (NGS) methods.

SECONDARY OUTCOMES:
Overall survival (OS) (Phase II) | From randomization to death due to any cause, or censored at the date last known alive, assessed up to 10 years
  OS distributions will be estimated using Kaplan-Meier (KM) methods and compared between treatment arms with the log-rank test. Stratified cox proportional hazards regression will produce a treatment hazard ratio estimate. Median OS by treatment arm with 95% confidence intervals will be reported.
Progression-free survival (PFS) (Phase II) | From randomization until the earlier of progression or death due to any cause, or censored at date of last disease evaluation, assessed up to 10 years
  PFS distributions will be estimated using KM methods and compared between treatment arms with the log-rank test. Stratified cox proportional hazards regression will produce a treatment hazard ratio estimate. Median PFS by treatment arm with 95% confidence intervals will be reported.
Best response (Phase II) | Up to cycle 8
  Will be based on standard IMWG criteria. Response will be tabulated by category. Response rates of very good partial response or better will be compared using the Fisher's exact test.
Time to progression (TTP) (Phase II) | From randomization to progression, or censored at the date of last disease evaluation, assessed up to 10 years
  TTP in each arm will be estimated using Kaplan-Meier methods and compared between arms with the log-rank test.
Incidence of adverse events (Phase II) | Up to 10 years
  Will be assessed per Common Terminology Criteria for Adverse Events version 5.0. Will compare worst grade 3 or higher non-hematologic and overall treatment-related toxicity rates between arms using the Fisher's exact test.

OTHER OUTCOMES:
Duration of treatment (Phase II) | From time of randomization to date off treatment, or censored at date of last treatment, assessed up to 10 years
  Treatment duration in each arm based on submission of the off-treatment case report form will be estimated using Kaplan-Meier methods and compared between arms with the log-rank test.
Cumulative dose (Phase II) | Up to 10 years
  Defined as the sum of all doses taken across all cycles. Descriptive statistics will be used to assess exposure to all drugs separately based on calculations for cumulative dose, dose intensity, and relative dose intensity.
Dose intensity (Phase II) | Up to 10 years
  Calculated as cumulative dose received divided by treatment duration. Descriptive statistics will be used to assess exposure to all drugs separately based on calculations for cumulative dose, dose intensity, and relative dose intensity.
Relative dose intensity (Phase II) | Up to 10 years
  Calculated as the dose intensity divided by planned dose intensity. Descriptive statistics will be used to assess exposure to all drugs separately based on calculations for cumulative dose, dose intensity, and relative dose intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Thompson, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (3):
- United States (3):
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm